CLINICAL TRIAL: NCT04707898
Title: Clinical Evaluation of Different Solvent-based Universal Adhesive Systems in Non-carious Cervical Lesions.
Brief Title: Clinical Evaluation of Different Universal Adhesive Systems in Non-carious Cervical Lesions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gulsah YENIER, Assist.Prof., Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/37-Rev/2
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Non-carious Cervical Lesions
Keywords: universal adhesive, non-carious lesions, randomized clinical trial

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Single Bond Universal (Experimental): Single Bond Universal adhesive system with selective-etch approach following the manufacturer's instruction
  Interventions: Device: Single Bond Universal
- Group G-Premio Bond (Experimental): G-Premio Bond Adhesive System with selective-etch approach following the manufacturer's instruction
  Interventions: Device: G-Premio Bond

INTERVENTIONS:
Device: Single Bond Universal — Adhesive system
  Arms: Group Single Bond Universal
Device: G-Premio Bond — Adhesive system
  Arms: Group G-Premio Bond

SUMMARY:
The aim of the study is to compare the performance of universal adhesives containing different-solvent-based in the restoration of non-carious cervical lesions (NCCLs).

DETAILED DESCRIPTION:
The study was approved by the Ethics Committee of the Istanbul University Faculty of Dentistry in accordance with protocol no. 2019/37-Rev/2. All participants will be informed about the study and will sign the written informed consent prior to the first treatment.

The tested materials are the universal adhesive systems: Single Bond Universal (3M ESPE, St. Paul, MN, USA) and G-Premio Bond (GC Corporation, Tokyo, Japan). Both adhesive systems will be used in selective-etch approach. All restorations will replaced by a single experienced dentist. In this study PASS 11 Software was used to calculate the sample size. At least 230 restorations (n=115) will be included for this study.

The patients will be given local anesthesia if required to prevent discomfort during the intervention. Prior to the restorative procedure the teeth will be cleaned with a pumice water slurry, using a rubber cup. The walls of the lesions are gently and superficially roughened using a round coarse diamond bur before adhesive procedures. Isolation of the tooth will be achieved by the use of cotton rolls and a saliva aspirator, a retraction cord (Ultrapak, Ultradent Products, Inc., South Jordan, USA). Both adhesives will be applied in manufacturer' s instructions with random order, by which the first randomly selected adhesive will be used to restore the tooth with the lowest tooth number (according to the FDI system), and the alternative adhesive will be used for the tooth with the second lowest tooth number. This method will be used for every other tooth requiring a cervical restoration. After adhesive procedures, resin composite will be placed and each increment light cured for 20 seconds (Elipar S10, 3M ESPE, St.Paul, MN, USA). The restorations are then finished and polished.

Restorations will be assessed 7 days after placement (baseline) and after 6, 12, 18, and 24months. Clinical examination will be performed by two blinded examiners, who were not involved in the treatments. Each restoration will be evaluated clinically using a dental loupe according to FDI World Dental Federation criteria. Three main groups- esthetic, functional, biological properties- and their sub-categorizes of FDI World Dental Federation criteria will be scored on a scale of 1 to 5.

Esthetic properties: Surface lustre, surface staining, marginal staining, color match and translucency, esthetical anatomical form

Functional properties: Fracture of material and retention, marginal adaptation, wear, approximal anatomical form, patient's view.

Biological properties: Post-operative sensitivity, recurrence of caries, erosion, abfraction, tooth integrity, periodontal response, adjacent mucosa, oral and general health.

Statistical analysis will be performed using IBM SPSS V23 Software. The data is analyzed with Chi- Square, Friedman Test, Bonferroni Test adjustment, Wilcoxon Tests (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Participant age should be 18-65 years.
* Good general health condition
* Good oral hygiene
* Should have at least 4 noncarious cervical lesion
* Must not have rampant caries
* At least 20 teeth in occlusion

Exclusion Criteria:

* Serious medical problems, allergies to product ingredients
* Poor oral hygiene
* Severe periodontal problems
* Caries or restorative treatment on teeth included in the study
* Parafunctional behavior
* Abutment of tested teeth to a removable prosthesis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
FDI World Dental Federation criteria | 24-months
  Retention and marginal adaptation

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University Faculty of Dentistry, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Landuyt KL, Peumans M, Fieuws S, De Munck J, Cardoso MV, Ermis RB, Lambrechts P, Van Meerbeek B. A randomized controlled clinical trial of a HEMA-free all-in-one adhesive in non-carious cervical lesions at 1 year. J Dent. 2008 Oct;36(10):847-55. doi: 10.1016/j.jdent.2008.06.005. Epub 2008 Jul 25. PMID 18656295
- [Background] Ermis RB, Van Landuyt KL, Cardoso MV, De Munck J, Van Meerbeek B, Peumans M. Clinical effectiveness of a one-step self-etch adhesive in non-carious cervical lesions at 2 years. Clin Oral Investig. 2012 Jun;16(3):889-97. doi: 10.1007/s00784-011-0565-4. Epub 2011 May 21. PMID 21603966
- [Background] Moretto SG, Russo EM, Carvalho RC, De Munck J, Van Landuyt K, Peumans M, Van Meerbeek B, Cardoso MV. 3-year clinical effectiveness of one-step adhesives in non-carious cervical lesions. J Dent. 2013 Aug;41(8):675-82. doi: 10.1016/j.jdent.2013.05.016. Epub 2013 Jun 6. PMID 23747824
- [Background] Lawson NC, Robles A, Fu CC, Lin CP, Sawlani K, Burgess JO. Two-year clinical trial of a universal adhesive in total-etch and self-etch mode in non-carious cervical lesions. J Dent. 2015 Oct;43(10):1229-34. doi: 10.1016/j.jdent.2015.07.009. Epub 2015 Jul 29. PMID 26231300
- [Background] Hafer M, Jentsch H, Haak R, Schneider H. A three-year clinical evaluation of a one-step self-etch and a two-step etch-and-rinse adhesive in non-carious cervical lesions. J Dent. 2015 Mar;43(3):350-61. doi: 10.1016/j.jdent.2014.12.009. Epub 2014 Dec 23. PMID 25541248
- [Background] Szesz A, Parreiras S, Reis A, Loguercio A. Selective enamel etching in cervical lesions for self-etch adhesives: A systematic review and meta-analysis. J Dent. 2016 Oct;53:1-11. doi: 10.1016/j.jdent.2016.05.009. Epub 2016 Jul 2. PMID 27381814
- [Derived] Yurdaguven GY, Dogruer I, Cam M, Ulukapi H, Aykor AA. Clinical evaluation of different solvent type and HEMA-content of universal adhesive systems in non-carious cervical lesions: a two-year double-blind split-mouth randomized clinical trial. BMC Oral Health. 2025 Oct 22;25(1):1661. doi: 10.1186/s12903-025-07081-0. PMID 41126209